CLINICAL TRIAL: NCT02127229
Title: The Impact of Cost Itemization on Resource Utilization With ERCP
Brief Title: Cost Analysis for Endoscopic Retrograde Cholangiopancreatography (ERCP)
Acronym: ERCP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled; study inactivated
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 574462
Record Dates: First submitted 2014-03-04; First posted 2014-04-30 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Biliary Obstruction
Keywords: endoscopic retrograde cholangiopancreatography; disposable accessory cost; endoscopy cost analysis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blinded observation of ERCP (No Intervention): Blind observation of disposable accessories use.
- Endoscopist informed of cost per procedure (Experimental): Endoscopists informed following each ERCP.
  Interventions: Procedure: Endoscopist informed of cost per procedure

INTERVENTIONS:
Procedure: Endoscopist informed of cost per procedure — Following each procedure, endoscopists will get a cost report regarding the amount spent on disposable accessories.
  Arms: Endoscopist informed of cost per procedure

SUMMARY:
The purpose of the study is to determine if endoscopist notification of accessory cost results in altered resource utilization related to the total cost and number of accessories used in ERCP.

This study will be a prospective cost--analysis study. Only chart review of PHI removed records will be used. The only intervention used is that endoscopists will be made aware of the cost of accessories used in the second phase of the study following each ERCP.

The investigators are in an era of increased medical cost consciousness. Medical education and post--graduate education incorporates cost savings and appropriate diagnostic test selection based on expense as one aspects of the decision process. This era now focuses on what is best for the patient with the understanding that the cost to the patient and cost to the overall health care system matters. Not only is this apart of postgraduate training but now being implemented as part of Medicare reimbursement to provide low cost and high quality care. Incidence of pancreatic and biliary disease is increasing. ERCP is a vital tool for therapeutic intervention. The costs of these procedures, to both patients and hospitals, have caused some to question the amount of accessories used as well as the poor reimbursement provided by Medicare and insurers. Studies have indicated that hospitals actually lose money with each ERCP used and their use is being limited many times to tertiary care centers.

DETAILED DESCRIPTION:
This study is a prospective cost-identification analysis of accessories used during the ERCP. The study will be conducted in two phases. Each phase will include at least 71 ERCP procedures. All consecutive patients undergoing ERCP will be included. For the first phase of the study the physicians performing the procedure will not be made aware of the study and also will not be briefed at the end of the procedure with the number of accessories used during the procedure and the dollar value of the accessories. For the second phase of the study, endoscopist will be briefed by the endoscopy manager after completion of each procedure about the total number of accessories used and the dollar value of the accessories used during the procedure.

During the study period, all gathered information will be deidentified but the procedure indication and whether it was successful or not will be collected. Only deidentified information will be collected. Endoscopists will not be aware of the study to avoid a Hawthorne effect. The endoscopists resource utilization is what is being studied. They will be debriefed at completion of protocol.

ERCP's requiring cholangioscopy (spyglass), stent removal alone, or just stent exchange will be excluded from the cost analysis, because of the atypical nature of the procedures and the number of accessories used during these procedures may not reflect the number of accessories used during a typical procedure. For both groups, if an endoscopic ultrasound is used for gaining biliary access it will be included in the cost analysis of this study. Both outpatient and inpatients will be included for both groups. All investigator patients will be excluded from the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult receiving ERCP at Endoscopy diagnostic center.

Exclusion Criteria:

* No stent removal or replacement procedures. EUS can only be used for intubation of bile duct. No spyglass will added to total cost.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of total cost of disposable accessories used for individual ERCP procedures | ERCP procedures will be observed for up to 3 months for each arms of study
  Two arms in the study. One arm is observation of blinding endoscopists and calculating cost of disposable accessories used while performing ERCP. The other arm will be the intervention group. Before the intervention period begins, advanced endoscopists will be informed that there cost is being monitored for each ERCP and the cost of disposable accessories. Following each ERCP during the intervention group, the endoscopists will be informed of the cost of that individual procedure based on disposable accessories.

SECONDARY OUTCOMES:
Cost identification of disposable accessory use in ERCP | ERCP procedures will be observed for up to 3 months for each arms of study
  Two arms in the study. One arm is observation of blinding endoscopists and calculating cost of disposable accessories used while performing ERCP. The other arm will be the intervention group. Before the intervention period begins, advanced endoscopists will be informed that there cost is being monitored for each ERCP and the cost of disposable accessories. Following each ERCP during the intervention group, the endoscopists will be informed of the cost of that individual procedure based on disposable accessories.

CONTACTS AND LOCATIONS:
Overall Officials: William Tierney, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Science Center, Oklahoma City, Oklahoma, United States